CLINICAL TRIAL: NCT00676468
Title: Comparative Effects of Fish Oil Supplementation and a Leukotriene Receptor Antagonist on EIB and Airway Inflammation in Asthma
Brief Title: Comparative Effects of Fish Oil Supplementation and a Montelukast on EIB and Airway Inflammation in Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Timothy D Mickleborough / Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-11765
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Asthma
Keywords: Asthma; Inflammation; Airway; Fish Oil; Singulair
MeSH Terms: conditions — Asthma; Inflammation | interventions — montelukast; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Active Montelukast + Fish Oil Placebo
  Interventions: Other: Active Montelukast + Fish Oil Placebo
- 2 (Other): Active Fish Oil + Montelukast Placebo
  Interventions: Other: Active Fish Oil + Montelukast Placebo
- 3 (Other): Active Montelukast + Active Fish Oil
  Interventions: Other: Active Montelukast + Active Fish Oil

INTERVENTIONS:
Other: Active Montelukast + Fish Oil Placebo — Montelukast (1 x 10 mg tablet) per day + 10 tablets of fish oil placebo (soy bean oil) per day for a duration of 3 weeks
  Other Names: Singulair (montelukast). Placebo (no brand name).
  Arms: 1
Other: Active Fish Oil + Montelukast Placebo — 10 tablets (3.2 g EPA + 2.0 g DHA) per day and 1 x 10 mg Montelukast Placebo tablet per day for a duration of 3 weeks.
  Other Names: Pro-Omega Fish Oil. Montelukast placebo (no brand name).
  Arms: 2
Other: Active Montelukast + Active Fish Oil — 1 x 10 mg Montelukast tablet per day and 10 tablets of active fish oil (3.2 g EPA + 2.0 g DHA) for a duration of 3 weeks.
  Other Names: Singulair (Montelukast) and Pro-Omega (Fish Oil).
  Arms: 3

SUMMARY:
Combining fish oil supplementation and Montelukast [a commonly used cyst LT1 receptor antagonist to treat exercise-induced bronchoconstriction (EIB)] will provide a greater antiinflammatory effect against developing EIB that either agent alone

DETAILED DESCRIPTION:
The aim of this study is to extend previous published findings that fish oil supplementation represents a beneficial treatment on exercise-induced bronchoconstriction (EIB). An important question is how dietary fish oil supplementation fits in with the available armamentarium [e.g., leukotriene (LT) modifiers] to decrease the expression of LTs, and whether fish oil supplementation may be additive, or used in its own right to block the EIB response. For example, it is possible that a combination of fish oil supplementation and a cyst LT1 receptor antagonist (LTRA) may provide a greater antiinflammatory effect against developing EIB that either agent alone.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrate a fall in post-exercise FEV1 of > 10% after dry air exercise challenge for the diagnosis of EIB and
* > 12% increase in FEV1 from the baseline value after the administration of a β2-agonist. However, if the bronchodilator response is < 12% increase in FEV1 from the baseline value then asthmatic subjects with EIB must further demonstrate
* A < 16.0 mg.ml-1 concentration of methacholine causing a 20% decrease in FEV1 (PC20)

Exclusion Criteria:

* Subjects will be excluded if they are pregnant
* Have a history of hyperlipidemia, hypertension, diabetes, bleeding disorders, delayed clotting time
* Taking aspirin medication and have a resting FEV1 less than 65% predicted.
* A complete blood count and urinary pregnancy tests will be conducted at the beginning of the study and subjects with a hematocrit < 35 will be excluded from participation in the study.
* In addition, subjects will also be excluded if they have a history of taking n-3 PUFA supplements or supplements with antioxidants above the levels recommended for Adequate Intake, or regularly consume more than one fish meal per week.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | 6 weeks

SECONDARY OUTCOMES:
Exhaled breathe condensate markers to measure airway inflammation | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Mickleborough, PhD, Study Director — Indiana University
Locations (1):
- Indiana University, Bloomington, Indiana, United States

REFERENCES:
- [Background] Mickleborough TD, Murray RL, Ionescu AA, Lindley MR. Fish oil supplementation reduces severity of exercise-induced bronchoconstriction in elite athletes. Am J Respir Crit Care Med. 2003 Nov 15;168(10):1181-9. doi: 10.1164/rccm.200303-373OC. Epub 2003 Aug 6. PMID 12904324
- [Background] Mickleborough TD, Lindley MR, Ionescu AA, Fly AD. Protective effect of fish oil supplementation on exercise-induced bronchoconstriction in asthma. Chest. 2006 Jan;129(1):39-49. doi: 10.1378/chest.129.1.39. PMID 16424411
- [Derived] Tecklenburg-Lund S, Mickleborough TD, Turner LA, Fly AD, Stager JM, Montgomery GS. Randomized controlled trial of fish oil and montelukast and their combination on airway inflammation and hyperpnea-induced bronchoconstriction. PLoS One. 2010 Oct 18;5(10):e13487. doi: 10.1371/journal.pone.0013487. PMID 20976161